CLINICAL TRIAL: NCT03364998
Title: Single Dose, Open Label, Randomized, Crossover Study in Subjects With Severe Hemophilia A Comparing Pharmacokinetic Parameters of BAY 94 9027 and Elocta
Brief Title: BAY94-9027 PK Study Comparing to Another Long Acting Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19096; 2017-003201-18 (EudraCT Number)
Record Dates: First submitted 2017-11-30; First posted 2017-12-07 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Intervention Model Description: Each subject will receive the two treatments. Pharmacokinetic samples will be collected from pre-dose until 120 hours after the end of the injection of the single dose in each treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BAY94-9027 and Elocta (Experimental): Subjects received two treatments: 60 IU/kg BAY94-9027 in the first period, followed by 60 IU/kg Elocta in the second period, with a washout period before each treatment
  Interventions: Drug: Damoctocog (Jivi, BAY94-9027); Drug: Elocta
- Elocta and BAY94-9027 (Experimental): Subjects received two treatments: 60 IU/kg Elocta in the first period, followed by 60 IU/kg BAY94-9027 in the second period, with a washout period before each treatment
  Interventions: Drug: Damoctocog (Jivi, BAY94-9027); Drug: Elocta

INTERVENTIONS:
Drug: Damoctocog (Jivi, BAY94-9027) — 60 international units (IU)/kg, given as a 10 minute injection, 1 dose
Drug: Elocta — 60 IU/kg, given as a 10 minute injection, 1 dose

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of BAY94-9027 and Elocta after intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 18 to 65 years.
* Subjects with Severe Hemophilia A with a documented plasma FVIII level of < 1%
* ≥ 150 exposure days with FVIII concentrate(s) as supported by medical records

Exclusion Criteria:

* Evidence of current or past inhibitor antibody:
* History of any congenital or acquired coagulation disorders other than hemophilia A.
* Platelet count <75,000/mm*3.
* Abnormal renal function (serum creatinine >2 x the upper limit of the normal range).
* Active liver disease verified by medical history or persistently elevated alanine aminotransferase or aspartate aminotransferase >5 x the upper limit of the normal range or severe liver disease as evidenced by, but not limited to any of the following: International Normalized Ratio >1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
AUC from time 0 to the last data point | Pre-Dose and up to 120 hours post dose
  Area under the concentration time profile curve.

CONTACTS AND LOCATIONS:
Locations (1):
- SHATHD Spec. Hospi. for Active Treatm. of Haematol. Dis. EAD, Sofia, Bulgaria

REFERENCES:
- [Derived] Shah A, Solms A, Wiegmann S, Ahsman M, Berntorp E, Tiede A, Iorio A, Mancuso ME, Zhivkov T, Lissitchkov T. Direct comparison of two extended-half-life recombinant FVIII products: a randomized, crossover pharmacokinetic study in patients with severe hemophilia A. Ann Hematol. 2019 Sep;98(9):2035-2044. doi: 10.1007/s00277-019-03747-2. Epub 2019 Jun 24. PMID 31236667
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/